CLINICAL TRIAL: NCT01939119
Title: Examination of the Body-fluid Balance in Patients With Retinal Vascular Occlusion Before and During Hemodilution and the Influence of Drinking Habits on the Degree of Body Hydration
Brief Title: Body-fluid Balance and Drinking Habits in Patients With Retinal Vascular Occlusion
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Technische Universität Dresden (Other)
Responsible Party: Principal Investigator, Dr. med. Evelyn Voigt, Dr. med., Technische Universität Dresden
Other Study IDs: VascOcclusion/Drinking2013
Record Dates: First submitted 2013-09-03; First posted 2013-09-11 (Estimated); Last update posted 2013-09-11 (Estimated); Status verified 2013-09

CONDITIONS: Dehydration; Retinal Vascular Occlusion
Keywords: retinal vascular occlusion; drinking habits; body hydration; body-fluid balance
MeSH Terms: conditions — Dehydration

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- retinal vascular occlusion: Patients with retinal vascular occlusion undergo a hematocrit dependent 5 day hemodilution

SUMMARY:
The purpose of this study is to examine the body-fluid balance in patients with retinal vascular occlusion and the influence of drinking habits and hemodilution on the degree of body hydration.

DETAILED DESCRIPTION:
Patients with retinal vascular occlusion who are hospitalized for hemodilution and cardiovascular risk assessment are asked to report their drinking habits. Hydration status before and during hemodilution is assessed with a body-fluid analyzing scale.

ELIGIBILITY:
Inclusion Criteria:

* informed consent
* age over 18 years

Exclusion Criteria:

* age under 18 years
* hypertensive urgency
* myocardial infarction < 4 weeks ago, chest pain
* heart rhythm disorders, high degree valvular defects
* pacemaker, defibrillator
* peripheral arterial occlusive disease
* end stage renal disease
* acute hepatitis, chronic inflammatory intestinal disease
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with retinal vascular occlusion
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2013-01; Primary Completion 2013-10 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
changes in body-fluid balance | 1 week
  The influence of hemodilution on body-fluid balance in patients with retinal vascular occlusion is examined

SECONDARY OUTCOMES:
number of participants with dehydration | 1 week
  All patients are asked to fill in a questionnaire concerning their drinking habits (thirst, fluid intake). Patients body-fluid balance during hemodilution is measured with bioimpedance spectroscopy (Body Composition Monitor, Fresenius)

CONTACTS AND LOCATIONS:
Overall Officials: Lutz E Pillunat, MD, Study Director — University Eye Clinic Dresden
Locations (1):
- University Eye Clinic, Dresden, Germany/ Saxony, Germany